CLINICAL TRIAL: NCT05813392
Title: Digital Cognitive Behavioral Therapy for Insomnia (dCBT-I) for Chronic Insomnia in Breast Cancer Survivors, A Randomized Controlled Trial
Brief Title: Digital Cognitive Behavioral Therapy for Insomnia for Chronic Insomnia in Breast Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Shenzhen Zeen Health Technology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Jing MA, Pro., Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-376
Record Dates: First submitted 2022-12-17; First posted 2023-04-14 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Chronic Insomnia
Keywords: Insomnia; Cognitive Behaviour Therapy for insomnia; breast cancer
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The enrolled breast cancer survivors were randomized into two groups: the intervention group was the dCBT-I treatment group and the control group was the wait-for-treatment group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dCBT-I group (Experimental): The dCBT-I group will receive full self-help dCBT-I through a smartphone APP for 6 weeks.
  Interventions: Behavioral: Digital Cognitive Behavioral Therapy for Insomnia
- the wait-list group (No Intervention): The wait-list group will not receive dCBT-I, waiting for treatment.At the end of the 3-month follow-up, the decision whether to receive treatment will be made according to the participants' wishes.

INTERVENTIONS:
Behavioral: Digital Cognitive Behavioral Therapy for Insomnia — a full self-help digital cognitive behavioral therapy for Insomnia (dCBT-I) through a smartphone APP
  Arms: dCBT-I group

SUMMARY:
To explore the efficacy of dCBT-I therapy for chronic insomnia among breast cancer survivors in China, we propose to conduct a randomized, parallel controlled clinical study in breast cancer survivors using a smartphone Chinese application (app) "resleep". Breast cancer survivors with chronic insomnia were recruited from our Breast Disease Center and externally, with the waiting group as a parallel control and the dCBT-I treatment group as an intervention group, in a 1:1 sample size. Intervention group (dCBT-I treatment group) will receive full self-help dCBT-I administered by smartphone APP for 6 weeks. The control group (waiting for treatment group) will not receive any additional interventions based on the original conventional treatment and will be followed up as planned, waiting for treatment.At the end of the 3-month follow-up, the decision to receive treatment was made according to the patient's wishes. The primary endpoint was the insomnia severity index (ISI) at the end of treatment and at 3 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Breast cancer diagnosed within 5 years
3. Stable disease at the end of acute treatment (surgery, radiotherapy, chemotherapy) while meeting: ≥ 1 month after surgery, ≥ 3 months after the end of last chemotherapy, and ≥ 3 months after the end of last radiotherapy if radiotherapy is required.
4. Satisfy the diagnostic criteria for chronic insomnia disorder according to the (International Classification of Sleep Disorders-the Third Edition, ICSD-3)[ and Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5): problem with falling asleep or maintaining sleep for ≥3 months (≥3 times per week) with impaired daytime functioning, despite the availability of sleep opportunities.
5. ISI score ≥12.
6. Other sleep or psychiatric disorders, if present, must be stable and require no medication.
7. Be proficient in the use of a cell phone application, and be comfortable reading, filling out the electronic questionnaire, communicating, and fully understanding the content.
8. Sign the informed consent form. -

Exclusion Criteria:

1. New breast cancer progression, recurrence, or metastasis within 3 months, requiring new radiotherapy or immunotherapy regimen
2. Expected survival <12 months due to all causes
3. Presence of any of the following conditions: Concurrent active cancer or malignancy that is being treated other than breast cancer, shift work, alcohol abuse, substance abuse, significant suicidal ideation, bipolar disorder, aggressive behavior, mania, schizophrenia.
4. Presence of a diagnosed significant physical illness that interferes with sleep, such as cranial disease or trauma, cancer pain, unstable angina, uncontrolled cardiac insufficiency and severe respiratory distress due to various causes, etc.
5. Current or previous treatment with cognitive behavior therapy for insomnia (CBT-I).
6. Not signed informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2023-08-29 (Actual); Primary Completion 2025-08-29 (Estimated); Study Completion 2026-08-29 (Estimated)

PRIMARY OUTCOMES:
The insomnia severity index (ISI) scores | immediately post-treatment
The insomnia severity index (ISI) scores | 3-months follow-up

SECONDARY OUTCOMES:
The insomnia severity index (ISI) scores | 6-months follow-up
Online sleep diary measures | up to 6-months follow-up
  Online sleep diary measures（total sleep time, sleep efficiency, sleep latency, numbers and duration of awakenings during sleep)

OTHER OUTCOMES:
Generalized Anxiety Scale (GAD-7) | up to 6-months follow-up
  The GAD-7 is a simple and reliable anxiety screening tool. There are a total of seven questions with a score of 0-3 for each question. The total score provides a possible score from 0-21. A score of 10 or greater indicates further evaluation is required.
Patient Health Questionnaire-9 (PHQ-9) | up to 6-months follow-up
  The PHQ-9 is a simple and validated self-assessment scale for depressive disorders, with good reliability and validity both as an aid to the diagnosis of depression and in the assessment of symptom severity. It has a total of nine items with a total score of 0-27.
the Short-Form 12 Health Survey (SF-12) | up to 6-months follow-up
  The SF-12 is a simplified version of the quality of life questionnaire generated based on the SF-36 scale, consisting of 12 items, containing eight dimensions, and assessing an individual's perceived physical and mental health status. The scale is scored on a percentage scale, and after obtaining a crude score, it is converted using the standardized scoring method. It includes the SF-12 Physical Component Summary (PCS) and Mental Component Summary (MCS) scores. Higher scores indicate higher levels of quality of survival.
  7)The smart bracelet data (recording parameters such as bedtime, sleep duration, number of awakenings during sleep, wake-up time, and sleep quality)
Pittsburgh sleep quality index (PSQI) | up to 6-months follow-up
the Functional Assessment of Cancer Therapy-Breast plus Arm morbidity (FACT-B + 4) | up to 6-months follow-up
EORTC Quality of Life Questionnaire (QLQ)-30 | up to 6-months follow-up
  EORTC: The European Organization for Research and Treatment of Cancer; QOL-C30: Quality of Life Questionnaire Core 30.

CONTACTS AND LOCATIONS:
Locations (1):
- Jing Ma, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811